CLINICAL TRIAL: NCT01514045
Title: The Gastric Cancer Foundation: A Gastric Cancer Registry
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20285; SU-01172012-8987 (Other: Stanford University); GI0005 (Other: OnCore)
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer
Keywords: Quality of Life
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples with DNA Paraffin embedded tissue will be stored in the Stanford Tissue Bank for 100 years.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Gastric Cancer Registry will combine data acquired directly from patients with gastric cancer; with a family history of gastric cancer in a first or second degree relative; or persons with a known germline mutation in their CDH1 (E-Cadherin) gene via an online questionnaire with genomic data obtained from saliva, blood and tissue samples. The purpose of this registry is to gain better understanding of the causes of gastric cancer, both environmental and genetic; whether certain genomic data can predict outcomes of treatment and survival.

DETAILED DESCRIPTION:
Collect detailed clinical and epidemiological information on eligible patients via an online registry and a detailed patient questionnaire. Participants can opt in to contribute a blood or saliva sample and paraffin block samples from a previous gastric surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are eligible if they have a histologically proven gastric tumor including gastroesophageal tumors; OR they have a family history of gastric cancer in a first or second degree relative; OR persons with a known germline mutation in their CDH1 (E-Cadherin) gene.
2. 18 years of age or older
3. Adequate English proficiency to complete online consent and questionnaire. Spanish-language proficiency as an alternative to English-language proficiency.

Exclusion Criteria:

1. Under 18 years of age
2. No history of gastric cancer or gastric cancer in a family member or a known germline mutation in their CDH1 gene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified for recruitment either by the individual's treating physician or through information about the registry on the Gastric Cancer Fund website. Potential participants will be directed to the URL for the gastric cancer registry and asked to complete a brief registration form which will include eligibility questions.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-04; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Collect detailed clinical and epidemiological information on patients with gastric cancer; with a family history of gastric cancer in a first or second degree relative; or persons with a known germline mutation in their CDH1 (E-Cadherin) gene | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Hanlee P Ji, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States